CLINICAL TRIAL: NCT00747149
Title: 12-week, Open-label, Multi-center, Prospective Study Evaluating the Effect of Individualizing Starting Doses of Rosuvastatin According to Baseline LDL (Low Density Lipoprotein)-Cholesterol Levels on Achieving Cholesterol Targets in Type 2 Diabetic Patients
Brief Title: A Diabetes Study to Treat A Population Previously Not at Target
Acronym: ADAPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3560L00072
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Results first posted 2011-07-04 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin 1 (Experimental): titrated
  Interventions: Drug: Rosuvastatin
- Rosuvastatin 2 (Experimental): Non-titrated
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Oral
  Other Names: Crestor

SUMMARY:
This study will assess if customizing the start dose of rosuvastatin appropriate for the degree of LDL-C reduction required, would achieve LDL-C target of ≤ 2.0 mmol/L quickly with either no titration or just one titration step after 6 weeks of therapy in type 2 diabetic patients previously treated with another statin and not at LDL-C targets.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 diabetes
* Previously treated with a commonly accepted start dose of a statin for the last 4 weeks prior to study entry
* Fasting LDL-C concentration of > 2.0 mmol/L (and ≤ 5.0 mmol/L) (in the past 3 months)
* History of serum TG level of ≤ 4.6 mmol/l (in the past 3 months)

Exclusion Criteria:

* If currently receiving therapy with any statin at a dose higher than listed
* Rosuvastatin (current use)
* Fibrates, niacin or resins that was not discontinued a minimum of 2 months prior to enrolment.
* Type 1 diabetes; glycated haemoglobin (HbA1c) > 9.0%
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥ 1.5 × upper limit of normal (ULN) (in the past 2 months)
* Resting diastolic or systolic blood pressure of > 95 mmHg or > 180 mmHg, respectively (in the past 2 months)
* Unexplained serum creatine kinase (CK) level > 3 × ULN (in the past 2 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Meani, Study Director — AstraZeneca; David Lau, MD, Principal Investigator — Private Practice
Locations (84):
- Canada (84):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Red Deer, Alberta
  - Research Site, Spruce Grove, Alberta
  - Research Site, St. Albert, Alberta
  - Research Site, Chilliwack, British Columbia
  - Research Site, Coquitlam, British Columbia
  - Research Site, Delta, British Columbia
  - Research Site, Kelowna, British Columbia
  - Research Site, Maple Ridge, British Columbia
  - Research Site, Penticton, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Portage la Prairie, Manitoba
  - Research Site, Winnipeg, Manitoba
  - Research Site, Bathurst, New Brunswick
  - Research Site, Woodstock, New Brunswick
  - Research Site, Carbonear, Newfoundland and Labrador
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Kentville, Nova Scotia
  - Research Site, Pubnico, Nova Scotia
  - Research Site, Sydney Mines, Nova Scotia
  - Research Site, Truro, Nova Scotia
  - Research Site, Aylmer, Ontario
  - Research Site, Bolton, Ontario
  - Research Site, Chatham, Ontario
  - Research Site, Fort Erie, Ontario
  - Research Site, Georgetown, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Morrisburg, Ontario
  - Research Site, Nepean, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Saint Catherines, Ontario
  - Research Site, Scaborough, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Smith Falls, Ontario
  - Research Site, St. Catharines, Ontario
  - Research Site, Thornhill, Ontario
  - Research Site, Thorold, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Welland, Ontario
  - Research Site, Willowdale, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Woodstock, Ontario
  - Research Site, Charlottetown, Prince Edward Island
  - Research Site, Kensington, Prince Edward Island
  - Research Site, Montague, Prince Edward Island
  - Research Site, Anjou, Quebec
  - Research Site, Dolbeau-Mistassini, Quebec
  - Research Site, Drummondville, Quebec
  - Research Site, Forestville, Quebec
  - Research Site, Gatineau, Quebec
  - Research Site, Joliette, Quebec
  - Research Site, L'Ile Perrot, Quebec
  - Research Site, La Sarre, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Roberval, Quebec
  - Research Site, Roxton Pond, Quebec
  - Research Site, Saint-bruno-lac-saint-jean, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saint-Léonard, Quebec
  - Research Site, Saint-Marc-des-Carrieres, Quebec
  - Research Site, Saint-Pie, Quebec
  - Research Site, Sainte Gedeon-de-beauce, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Thetford-Mines, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Moose Jaw, Saskatchewan
  - Research Site, Porcupine Plain, Saskatchewan
  - Research Site, Saskatoon, Saskatchewan
  - Research Site, Yorkton, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1044 patients (adult male and non-pregnant females) were enrolled at 122 Canadian family practice sites between May 2008 and May 2009. Out of these, only 598 patients were allocated to treatment. The remaining 446 did not receive treatment as they did not fulfill the inclusion/exclusion criteria.
Pre-assignment Details: Following enrolment, at Visit 1 the patients' Low Density Lipoprotein Cholesterol (LDL-C) value was baselined. If LDL-C value from Visit 1 was > 2.00, but ≤ 2.50 mmol/L: patients received Rosuvastatin (RSV)10 mg under the RSV 10 mg arm. If LDL-C value from Visit 1 was > 2.50 mmol/L: patients received Rosuvastatin 20 mg under the RSV 20 mg arm.
Groups:
- Rosuvastatin Titrated: 10 mg rosuvastatin (RSV) as initial dose followed by 20 mg RSV as titrated dose or 20 mg rosuvastatin (RSV) as initial dose followed by 40 mg RSV as titrated dose
- Rosuvastatin Non-titrated: 10 mg RSV or 20 mg RSV
Period: Overall Study
Arm/Group | Rosuvastatin Titrated | Rosuvastatin Non-titrated
Started | 154 | 444
Completed | 153 | 401
Not Completed | 1 | 43
Not completed — Adverse Event | 0 | 15
Not completed — Lost to Follow-up | 0 | 10
Not completed — Withdrawal by Subject | 0 | 6
Not completed — Did not receive treatment | 0 | 1
Not completed — Incorrect enrollment | 0 | 6
Not completed — Severe non-compliance to protocol | 0 | 1
Not completed — Not reported | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Rosuvastatin 10 mg (Initial): 10 mg rosuvastatin (RSV) as initial dose
- Rosuvastatin 20 mg (Initial): 20 mg RSV as initial dose
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin 10 mg (Initial) | Rosuvastatin 20 mg (Initial) | Total
Number analyzed (Participants) | 319 | 279 | 598
Age Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (10.9) | 62.6 (10.5) | 62.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 145 | 295
  Male | 169 | 134 | 303
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 288 | 245 | 533
  Black/African American | 5 | 7 | 12
  Asian | 22 | 17 | 39
  Other | 4 | 10 | 14
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2]
  BMI | 32.50 (6.89) | 32.27 (6.72) | 32.39 (6.81)
Waistline circumference [Mean (Standard Deviation); unit: cm] | 106.7 (14.9) | 106.7 (15.9) | 106.7 (15.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Canadian Low Density Lipoprotein Cholesterol (LDL-C) Target Goals (i.e. LDL-C ≤ 2.0 mmol/L) After 12 Weeks of Rosuvastatin Therapy
Description: The number of subjects achieving Canadian Low density lipoprotein cholesterol (LDL-C) target goals (i.e. LDL-C ≤ 2.0 mmol/L) over the total number subjects treated after 12 weeks of rosuvastatin therapy multiplied by 100
Time Frame: 12 Weeks
Measure: Mean (95% Confidence Interval); unit: Percentage
Groups:
- Rosuvastatin 10 mg (Initial); Rosuvastatin 20 mg (Initial); Rosuvastatin 20 mg (Titrated); Rosuvastatin 40 mg (Titrated): At visit 1, LDL C level was measured. At visit 2, subjects received treatments with rosuvastatin 10 mg or 20 mg based on their visit 1 LDLC level. At visit 3 (6 weeks after visit 2) LDLC values was measured again and patients were titrated to the next highest dose of rosuvastatin if they had not reached target level of LDLC. Hence, 4 arms are listed, subjects who started on 10 mg could be on 10mg, 20mg by the end of the study and those subjects who started on 20mg could be on 20mg or 40 mg at the end of the study.
Arm/Group | Rosuvastatin 10 mg (Initial) | Rosuvastatin 20 mg (Initial) | Rosuvastatin 20 mg (Titrated) | Rosuvastatin 40 mg (Titrated)
Number analyzed (Participants) | 225 | 176 | 75 | 78
Percentage | 87 (82) [82 to 91] | 87 (81) [81 to 91] | 76 (65) [65 to 84] | 63 (52) [52 to 73]

2. Secondary Outcome: Percentage of Subjects Achieving Total Cholesterol (TC)/ High-density Lipoprotein Cholesterol (HDLC) Ratio (i.e. TC/HDL < 4.0 mmol/L) at 6 and 12 Weeks of Treatment
Description: Proportion of subjects achieving total cholesterol (TC)/ High-density lipoprotein cholesterol (HDLC) ratio (i.e. TC/HDL < 4.0 mmol/L) at 6 and 12 weeks of treatment
Time Frame: 6 and 12 Weeks
Reporting Status: Not Posted
Measure: Mean (95% Confidence Interval); unit: Percentage of participants

3. Secondary Outcome: Mean Percent Change in Total Cholesterol (TC), Low Density Lipoprotein Cholesterol (LDL-C), High-density Lipoprotein Cholesterol (HDLC) , TC/HDL-C Ratio, Non-HDL-C, Triglycerides and Apolipoprotein B (ApoB) /Apolipoprotein A1 (ApoA-1) Ratio
Time Frame: 6 and 12 Weeks
Reporting Status: Not Posted
Measure: Mean (95% Confidence Interval); unit: Percentage

4. Secondary Outcome: Mean High Sensitivity C-reactive Protein (hsCRP) Value at Week 6 and 12
Time Frame: 6 and 12 Weeks
Reporting Status: Not Posted
Measure: Mean (95% Confidence Interval); unit: value mg/L

5. Secondary Outcome: Incidence of Adverse Events and Abnormal Laboratory Values After 12 Weeks of Therapy
Time Frame: 6 and 12 Weeks
Reporting Status: Not Posted
Measure: Number; unit: Participants

ADVERSE EVENTS:
Groups:
- Rosuvastatin 10 mg (Continued, Non-titrated): 10 mg RSV as a continued, non-titrated dose
- Rosuvastatin 20 mg (Continued, Non-titrated): 20 mg RSV as continued, non-titrated dose
- Rosuvastatin 20 mg (Titrated); Rosuvastatin 40 mg (Titrated): 20 mg RSV as titrated dose
Arm/Group | Rosuvastatin 10 mg (Initial) | Rosuvastatin 10 mg (Continued, Non-titrated) | Rosuvastatin 20 mg (Initial) | Rosuvastatin 20 mg (Continued, Non-titrated) | Rosuvastatin 20 mg (Titrated) | Rosuvastatin 40 mg (Titrated)
Serious Adverse Events (participants affected / at risk) | 4/319 | 2/232 | 0/279 | 0/182 | 1/75 | 1/78
Other Adverse Events (participants affected / at risk) | 14/319 | 4/232 | 9/279 | 3/182 | 2/75 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 10 mg (Initial) (N=319) | Rosuvastatin 10 mg (Continued, Non-titrated) (N=232) | Rosuvastatin 20 mg (Initial) (N=279) | Rosuvastatin 20 mg (Continued, Non-titrated) (N=182) | Rosuvastatin 20 mg (Titrated) (N=75) | Rosuvastatin 40 mg (Titrated) (N=78)
Labyrinthitis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chemical Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Aortic Aneurysm Rupture (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 10 mg (Initial) (N=319) | Rosuvastatin 10 mg (Continued, Non-titrated) (N=232) | Rosuvastatin 20 mg (Initial) (N=279) | Rosuvastatin 20 mg (Continued, Non-titrated) (N=182) | Rosuvastatin 20 mg (Titrated) (N=75) | Rosuvastatin 40 mg (Titrated) (N=78)
Constipation (Gastrointestinal disorders) | 5 | 0 | 6 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 2 | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca shall have a period of 30 days from receipt of the proposed final manuscript for any publication or other disclosure to review it and may within such time require that submission for publication or disclosure of the manuscript be delayed in order for AstraZeneca to file patent applications.